CLINICAL TRIAL: NCT05523947
Title: A Phase 1/2, Open-label, Multicenter, First-in-Human Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Anti-tumor Activity of YH32367 in Patients With HER2-Positive Locally Advanced or Metastatic Solid Tumors
Brief Title: Clinical Trial of YH32367 in Patients With HER2 Positive Locally Advanced or Metastatic Solid Tumor
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YH32367-101
Record Dates: First submitted 2022-08-24; First posted 2022-09-01 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2026-01

CONDITIONS: HER2-Positive Solid Tumor
Keywords: YH32367; HER2/4-1BB bispecific antibody; Solid tumor; Breast cancer; Gastric cancer; HER2-positive; Biliary tract cancer
MeSH Terms: conditions — Breast Neoplasms; Stomach Neoplasms; Biliary Tract Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- YH32367 (Experimental): Dose Escalation Part: 8 Cohorts. In Dose Escalation part, patients are assigned to receive YH32367 at a starting dose and the dose being escalated/de-escalated in adjacent dose cohorts.
  Dose Expansion Part: 2 Cohorts (Cohort 1: Biliary tract cancer, Cohort 2: Solid tumors). Dose Expansion part will consist of multiple cohorts in patients who were treated with at least 1 prior gemcitabine- and/or cisplatin-based therapy, HER2 positive biliary tract cancer(Cohort 1); in patients who were treated with all available standard therapies and have no available options, HER2 positive solid tumor malignancies other than breast and gastric or gastroesophageal junction adenocarcinoma and biliary tract cancer(Cohort 2).
  Interventions: Drug: YH32367

INTERVENTIONS:
Drug: YH32367 — Dose Escalation Part: 8 Cohorts. In this part, approximately 30 patients will be enrolled and patients are assigned to receive YH32367 at a starting dose and the dose being escalated/de-escalated in adjacent dose cohorts will be up to Dose level 8.
  Dose Expansion Part: 2 Cohorts(Cohort 1: Biliary tract cancer, Cohort 2: Solid tumors). The part will consist of multiple cohorts in patients who were treated with at least 1 prior gemcitabine- and/or cisplatin-based therapy, HER2 positive biliary tract cancer(Cohort 1); in patients who were treated with all available standard therapies and have no available options, HER2 positive solid tumor malignancies other than breast and gastric or gastroesophageal junction adenocarcinoma and biliary tract cancer(Cohort 2). Each cohort will enroll 65 and 40 patients, respectively.

SUMMARY:
This first-in-human study will be counducted to evaluate the safety, tolerability, pharmacokinetics (PK) and anti-tumor activity of YH32367 in Patients with HER2-Positive Locally Advanced or Metastatic Solid Tumors.

DETAILED DESCRIPTION:
YH32367, a novel HER2/4-1BB bispecific antibody (BsAb), simultaneously targets HER2 and h4-1BB and binds to both targets. YH32367 exhibits a strong 4-1BB signal activation as well as blocking of HER2 signaling in HER2-expressing tumor cells. YH32367 stimulates IFN-γ secretion from T cells and thereby induces tumor cells lysis.

This is a Phase 1/2, open-label, multicenter, first-in-human study of YH32367. This 2-part study will include both a Dose Escalation part, to identify the Maximum Tolerated Dose (MTD) and/or two dose levels for RP2D selection, and a Dose Expansion part, to determine RP2D and to confirm the safety, tolerability and efficacy of YH32367 at the RP2D.

ELIGIBILITY:
Inclusion Criteria:

[Dose Escalation Part]

* Pathologically confirmed HER2-positive
* Mandatory provision of tumor tissue sample

[Dose Expansion Part]

* Patients who have at least one measurable lesion
* Mandatory provision of tumor tissue sample

  1. Cohort 1: Pathologically confirmed HER2-positive biliary tract cancer
  2. Cohort 2: Pathologically confirmed HER2-positive metastatic solid tumor malignancy other than breast and gastric or gastroesophageal junction adenocarcinoma and biliary tract cancer

Exclusion Criteria:

* Uncontrolled central nervous system (CNS) metastases
* Spinal cord compression
* Carcinomatous meningitis
* Acute coronary syndromes
* Heart failure
* Interstitial lung disease (ILD)
* Pneumonitis
* History of a second primary cancer
* Human immunodeficiency virus (HIV)
* Active chronic hepatitis B
* Hepatitis C
* Systemic steroid therapy
* Autoimmune disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Estimated)
Dates: Start 2022-08-26 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Treatment-emergent adverse events (TEAEs) up to Day 21 | in dose escalation part, an average of 21 days
  To assess the safety and tolerability of YH32367
Objective Response Rate (ORR) | through dose expansion part completion, approximately 2.5 year
  To assess the ORR of YH32367 at the recommended Phase 2 dose (RP2D) according to RECIST v1.1 by blinded independent central reviews (BICR)

SECONDARY OUTCOMES:
Area under the serum concentration-time curve from time 0 to the last quantifiable concentration (AUClast) | up to 66 weeks
  To characterize the PK of YH32367
maximum observed serum concentration (Cmax) | up to 66 weeks
  To characterize the PK of YH32367
time to reach Cmax (Tmax) | up to 66 weeks
  To characterize the PK of YH32367
Presence and characterization of YH32367 ADA in serum including titer of ADA and neutralizing antibodies | through study completion, approximately 3.5 year
  To explore the immunogenicity of YH32367
Objective Response Rate (ORR) | through study completion, approximately 3.5 year
  To assess the anti-tumor efficacy according to RECIST v1.1 by Investigator assessment
Duration of Response (DoR) | through study completion, approximately 3.5 year
  To assess the anti-tumor efficacy according to RECIST v1.1 by Investigator assessment
Disease Control Rate (DCR) | through study completion, approximately 3.5 year
  To assess the anti-tumor efficacy according to RECIST v1.1 by Investigator assessment
Depth of Response | through study completion, approximately 3.5 year
  To assess the anti-tumor efficacy according to RECIST v1.1 by Investigator assessment
Time to Response | through study completion, approximately 3.5 year
  To assess the anti-tumor efficacy according to RECIST v1.1 by Investigator assessment
Progression-free survival (PFS) | through study completion, approximately 3.5 year
  To assess the anti-tumor efficacy according to RECIST v1.1 by Investigator assessment
TEAEs | through dose expansion part completion, approximately 2.5 year
  To assess the safety and tolerability of YH32367 at the RP2D
Overall Survival (OS) | through study completion, approximately 3.5 year
  To assess overall survival of YH32367

OTHER OUTCOMES:
Immune ORR (iORR) | through study completion, approximately 3.5 year
  To assess the immune-related efficacy according to iRECIST by Investigator assessment
Immune Duration of Response (iDOR) | through study completion, approximately 3.5 year
  To assess the immune-related efficacy according to iRECIST by Investigator assessment
Immune PFS (iPFS) | through study completion, approximately 3.5 year
  To assess the immune-related efficacy according to iRECIST by Investigator assessment

CONTACTS AND LOCATIONS:
Overall Officials: Hyejin Choi, Principal Investigator — Severance Hospital; Kyu-pyo Kim, Principal Investigator — Asan Medical Center; Do-Youn Oh, Principal Investigator — Seoul National University Hospital; Joon Oh Park, Principal Investigator — Samsung Medical Center; Ganessan Kichenadasse, Principal Investigator — Southern Oncology Clinical Research Unit; Jennifer Man, Principal Investigator — Blacktown Hospital; Arlene Chan, Principal Investigator — Breast Cancer Research Centre WA; Ju Won Kim, Principal Investigator — Korea University Anam Hospital; Myung Ah Lee, Principal Investigator — The Catholic University of Korea, St. Mary's hospital; Hongjae Chon, Principal Investigator — CHA Bundang Medical Center; Niall Tebbutt, Principal Investigator — Austin Health; Jung Hun Kang, Principal Investigator — Gyeongsang National University Hospital; Seok Yun Kang, Principal Investigator — Ajou University School of Medicine; Hyung Soon Park, Principal Investigator — Catholic University of Korea St. Vincent's Hospital; Ji Hong Bae, Principal Investigator — Gachon Gil University Medical Center; Cheol Kyung Sin, Principal Investigator — Ulsan University Hospital; Hae Seong Park, Principal Investigator — Dana-Farber Cancer Institute; Thatcher Heumman, Principal Investigator — Vanderbilt-Ingram Cancer Center; Hongsik Kim, Principal Investigator — Chungbuk National University Hospital
Locations (19):
- United States (2):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Vanderbilt Ingram Cancer Center, Nashville, Tennessee
- Australia (4):
  - Southern Oncology Clinical Research Unit, Adelaide
  - Austin Health, Melbourne
  - Breast Cancer Research Centre - WA, Perth
  - Blacktown Hospital, Sydney
- South Korea (13):
  - CHA Bundang Medical Center, Seongnam-si, Gyeonggi-do
  - Catholic University of Korea St. Vincent's Hospital, Suwon, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Gyeongsang National University Hospital, Jinju, Gyeongsangnam-do
  - Chungbuk National University Hospital, Cheongju-si, North Chungcheong
  - Gachon Gil University Medical Center, Incheon
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, St. Mary's hospital, Seoul
  - Ulsan University Hospital, Ulsan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (including data dictionaries) that underline the results reported in study-related publications will be made available during the period beginning 1 year and ending 5 years after all trial primary and secondary endpoints were assessed. Only requests from researchers who provide a methodologically sound proposal will be reviewed and approved by the sponsor. The analysis type should be in accordance with aims in the proposal approved by the sponsor. Proposals should be directed to andrew90@yuhan.co.kr.
  A summary of the study results will be posted in the publicly accessible database (i.e. clinicaltrials.gov) no later than 1 year after the study's primary completion date.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Beginning 1 year and ending 5 years after all trial endpoints were assessed
Access Criteria: Only requests from researchers who provide a methodologically sound proposal will be reviewed and approved by the sponsor. The analysis type should be in accordance with aims in the proposal approved by the sponsor. Proposals should be directed to andrew90@yuhan.co.kr.